CLINICAL TRIAL: NCT02561286
Title: Help Us, Save Us! HIV/STI Risk Reduction for Black Men Who Have Sex With Men
Brief Title: Being Responsible for Ourselves HIV Risk Reduction for Black MSM
Acronym: BRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 806708; R01MH079736 (NIH)
Record Dates: First submitted 2015-09-24; First posted 2015-09-28 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Human Immunodeficiency Virus Infection (HIV); Sexually Transmitted Disease (STD)
Keywords: Human immunodeficiency virus; Sexually transmitted disease; Men who have sex with men; African Americans; Behavioral intervention; Randomized controlled trial; Sexual behavior; Mediation analysis; Social cognitive theory; Theory of planned behavior
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases; Homosexuality; Sexual Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIV risk reduction (Experimental): BRO HIV Risk Reduction Intervention
  Interventions: Behavioral: BRO HIV Risk Reduction Intervention
- Health promotion control (Active Comparator): Health Promotion Intervention
  Interventions: Behavioral: Health Promotion Intervention

INTERVENTIONS:
Behavioral: BRO HIV Risk Reduction Intervention — BRO HIV Risk Reduction Intervention was designed to strengthen outcome expectancies supporting condom use and other sexual risk reduction strategies and skill and self-efficacy to use condoms and reduce sexual risk behaviors. It consisted of three 90-min one-on-one individual sessions implemented during 3 consecutive weeks by specially trained facilitators using standardized intervention manuals. Sessions 1 and 2 included take-home assignments that the participants reviewed at the subsequent session. The delivery of the intervention was tailored to the information that the participants provided during the sessions, including the context in which behaviors occurred and participants' motivation for the behaviors.
  Other Names: HIV Risk Reduction Intervention
  Arms: HIV risk reduction
Behavioral: Health Promotion Intervention — Health Promotion Intervention was designed to provide a control for "Hawthorne effects," reducing the likelihood that the HIV/STI risk-reduction intervention's effects could be attributed to non-specific features, including special attention. It focused on increasing physical activity and fruit-and-vegetable consumption and decreasing fat consumption to reduce the risk of chronic diseases, including heart disease, hypertension, stroke, diabetes, and certain cancers-leading causes of morbidity and mortality among African Americans It also consisted of three 90-min one-on-one individual sessions implemented during 3 consecutive weeks by specially trained facilitators using standardized intervention manuals.
  Other Names: Attention Control Intervention; BRO Health Promotion Intervention; Health Promotion Control
  Arms: Health promotion control

SUMMARY:
The incidence of HIV/AIDS among African American men who have sex with men (MSM) is alarming, and the public health response to this urgent situation has been hampered by a lack of sexual risk reduction interventions with solid evidence of efficacy in this population. Accordingly, the broad, long-term objective of the proposed research is to identify interventions to reduce the risk of sexually transmitted infection (STI) among African American MSM. This application seeks funds to develop and test the efficacy of a theory-based, contextually appropriate behavioral intervention to reduce sexual risk behavior among African American MSM. Intervention development will be guided by social cognitive theory, the theory of planned behavior, qualitative information from focus groups, and findings from a longitudinal survey of men from the study population. A one-on-one intervention will be utilized to address the specific prevention needs of each man and to allay participants' concerns about revealing their sexual involvement with men by virtue of participating in a group or workshop intervention. The study will utilize a randomized controlled trial design, with baseline, immediate post intervention, and 6 and 12 months post intervention assessments. The participants will be African American MSM who will be randomized to a one-on-one sexual risk reduction intervention or a one-on-one health promotion intervention that will serve as the control condition. The primary outcome is consistent condom use during anal and vaginal intercourse. The study will test whether the intervention increases the consistent use of condoms during anal intercourse, the primary outcome, whether it decreases other sexual risk behaviors, and whether social cognitive theory variables mediate the effects of the intervention on consistent condom use. This study will provide an urgently needed intervention to reduce the risk of HIV and other STIs in one of the highest risk populations in the United States.

DETAILED DESCRIPTION:
HIV/AIDS has had a devastating impact on African American MSM. Although African Americans represent only 13% of the US population, 49% of AIDS diagnoses in 2004 were in African Americans. That HIV/AIDS has taken an increasing toll on African American injection drug users and heterosexuals during the last decade is well documented. Nevertheless, MSM continue to account for the largest number of African Americans with HIV/AIDS. Through 2004, the MSM exposure category accounted for 37% of the cumulative AIDS cases in African American men, whereas injection drug use accounted for 31% and heterosexual transmission accounted for 10%. Consonant with these figures on HIV/AIDS cases, the HIV infection rates in several studies the Centers for Disease Control and Prevention (CDC) conducted on African American MSM have rivaled those found in many sub-Saharan African nations. For instance, a CDC 5-city study found that of the African American MSM who were tested for HIV, two-thirds were unaware of their status and 46% were HIV positive. Similarly, the 7-city CDC Young Men's Survey found an HIV prevalence rate of 32% in African American MSM. Interestingly, although African American MSM have relatively high HIV infection rates, evidence does not suggest that they engage in riskier sexual practices than do other MSM. This may mean that African American MSM are drawing their sexual partners from pools of people where HIV prevalence is relatively high, which underscores the urgency of targeting interventions to this population.

Quite apart from risk of HIV, African American MSM are at high risk for other STIs. The CDC MSM Prevalence Monitoring Project conducted in 9 US cities, in 1999 through 2004 found that the rates of gonorrhea and chlamydia were high in MSM, but especially high in African American MSM. In 2004, urethral gonorrhea positivity was 16% in African Americans, as compared with 11% in Whites, and 9% in Hispanics. The median urethral chlamydia positivity was 6% overall, but 9% in African Americans. To curb the HIV epidemic and the high rates of other STIs in African American MSM now, prevention efforts must be urgently undertaken.

Although several researchers have stressed the need for culturally appropriate prevention interventions targeting African American MSM, scant progress has been made toward the identification of such interventions. Ample evidence indicates that theory-based interventions can decrease sexual risk behavior among MSM. A meta-analysis 40 controlled studies of HIV prevention behavioral interventions for MSM found that the interventions reduced the amount of reported unprotected sex by as much as 27%, but revealed that the MSM populations at the highest risk, including African American MSM, have been underserved by intervention research. Consider, for example, Project EXPLORE, a large-scale multi-site controlled trial (RCT) that enrolled over 4,200 MSM and followed them for up to 4 years. Fewer than 7% of participants were African American, eligible African Americans were less likely to enroll in the trial than were eligible Whites, and African Americans were more likely to drop out. Another meta-analysis found that, of 33 HIV sexual risk reduction intervention trials on MSM, only 6 employed a sample that was at least a 10% African American. The insufficient number of rigorous intervention trials directed at African American MSM has hindered the ability to make definitive conclusions about how to combat men's attitudes and beliefs concerning sexual risk behavior and ultimately determine the effectiveness of HIV prevention strategies targeting African American MSM.

Reaching African American MSM may be particularly challenging because many African American MSM do not use traditional resources and organizations that serve gay men because they do not identify with White gay culture. In addition, African American MSM may also be difficult to reach within African American communities because they are often closeted and isolated due to real and perceived homophobia. That isolation, in turn, contributes to internalized repression of gay sexual identity, which may further isolate them from resources available to gay men. The investigators' approach to addressing the problem of reaching African American MSM is to develop an intervention that can be used by community-based organizations (CBOs) that already serve African American MSM. The investigators will create a Community Advisory Board that includes representatives of CBOs that serve African American MSM and representatives of the study population to advise them on the intervention design and other aspects of the trial. In addition, the investigators have held a focus group with representatives of CBOs that serve African Americans and have frequently consulted with them regarding their approach.

Reviews of the literature have suggested that there have been 3 basic approaches to the design of HIV/STI risk reduction programs aimed at MSM. One approach is to seek to reduce risk through the implementation of small group or workshop interventions. The second approach is through the use of community-level interventions. A third approach is the individual one-on-one intervention. All three approaches have merit and have reduced risk behavior among men in controlled trials. An advantage of the one-on-one is that it avoids the problem of men having to risk revealing that they have sex with other men in order to participate in the prevention program. There are added benefits of the one-on-one approach. It permits tailoring the intervention to the specific needs of the man. A recent meta-analysis has identified characteristics of effective HIV behavioral interventions for MSM. Efficacy was associated with interventions having more than one session, duration of 4 or more hours, and a time span of at least 3 weeks.

The Proposed Randomized Controlled Trial (RCT)

This study will test the efficacy of the Being Responsible for Ourselves (BRO) HIV Risk Reduction Intervention in increasing condom use and reducing other sexual risk behaviors among African American MSM in Philadelphia, where African Americans account for 70% of the reported cases of AIDS through June 2005. The study will use a RCT design, which is the most scientifically sound method for assessing the causal impact of interventions. An attention-matched control group, the Health Promotion Intervention, will provide controls for Hawthorne effects and special attention. Computer-generated random number sequences will be used to randomly assign participants to the intervention arms using concealment of allocation techniques designed to minimize bias in assignment. The biostatistician will generate the random assignments; the project director will implement the assignments. The study will also examine theoretical variables the intervention is designed to affect, which will permit mediation analyses addressing why the intervention is efficacious or not efficacious. This study, then, will provide an urgently needed intervention to help curb the alarmingly high incidence of HIV in urban, African American communities.

The BRO HIV Risk Reduction Intervention and the Health Promotion Intervention were developed based on social cognitive theory and the reasoned action approach, integrated with extensive formative research, including focus groups and pilot testing. Most relevant here are the social-cognitive-theory constructs of "outcome expectancy," beliefs about the consequences of a specific behavior, and "self-efficacy," people's confidence that they can execute a specific behavior; its emphasis on behavioral skills; and its methods for increasing skills, particularly practice with performance feedback (e.g., role-playing). The reasoned action approach is an extension of the theory of planned behavior, which itself is an extension of the theory of reasoned action. Most relevant here are the reasoned action approach's emphasis on the importance of salient beliefs, its notion that such beliefs may vary from population to population and from behavior to behavior, and its methods to identify such population-specific beliefs: namely, the use of qualitative research, including focus groups. By identifying and targeting a population's salient beliefs, an intervention can change those beliefs resulting in changes in the targeted behavior. The investigators utilized one-on-one interventions to allay concerns some African American MSM might have about revealing their sexual behavior with other men by virtue of participating in a group-based intervention, a concern expressed in the focus groups with African American MSM and with representatives of CBOs serving African American MSM.

Consistent with the reasoned action approach, the investigators conducted qualitative research, including 7 focus groups with African American MSM and 1 with representatives of CBOs that serve African American MSM, to ensure the intervention was tailored to the population. In addition, the investigators conducted 3 pilot tests of the interventions. The BRO HIV/STI risk-reduction intervention was designed to strengthen outcome expectancies expressed in focus groups with African American MSM, outcome expectancies that have been observed in other populations, including the hedonistic outcome expectancy that using condoms would not interfere with sexual enjoyment, the prevention outcome expectancy that using condoms prevents STIs, including HIV, and the self-evaluative outcome expectancy that using condoms would make the man feel good about himself. The intervention was designed to address aspects of self-efficacy identified in the focus groups, including technical-skill self-efficacy to use condoms correctly without interfering with sexual enjoyment, impulse-control self-efficacy to exercise the necessary control to use condoms even when sexually excited, under the influence of alcohol or drugs, or in the presence of other triggers for unsafe sex, and skills and self-efficacy to negotiate condom use with sexual partners. In addition, it was designed to increase knowledge regarding the risk of acquiring or transmitting HIV and other STIs, and perceived vulnerability to HIV infection or re-infection with a different strain of HIV.

Summary

In summary, African Americans have been disproportionately affected by the HIV epidemic. The prevalence of HIV infection among African American MSM is alarmingly high, paralleling rates observed in some countries in sub-Saharan Africa. For condoms to prevent the transmission of HIV/AIDS, they must be used correctly and consistently. Behavioral interventions have been found to be effective in reducing rates of sexual risk behaviors, but few have been conducted with African American MSM. This research seeks to answer the call for culturally appropriate interventions for high-risk subgroups of MSM. The primary hypothesis is that the BRO HIV Risk Reduction Intervention will increase the consistent use of condoms and decrease other sexual risk behaviors compared with the control group and that the intervention's effects on condom use with be mediated by variables from the social cognitive theory and the reasoned action approach.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Self-identified as black or African American
* Born a male
* Reported having anal intercourse with a man in the previous 90 days.

Exclusion Criteria:

* Reported having anal intercourse with only one main male partner in the past 90 days
* Participated in an HIV/STI risk-reduction intervention in the past 12 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 595 (Actual)
Dates: Start 2008-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Consistent (100%) condom use during anal and vaginal intercourse in the past 3 months | 6 and 12 months post-intervention
  Men who reported at least one intercourse act and whose number of reported protected acts equaled their number of acts were coded as practicing consistent condom use. Men who reported at least one intercourse act and whose reported number of protected acts was less than their number of acts were coded as not practicing consistent condom use.

SECONDARY OUTCOMES:
Receptive anal intercourse in the past 3 months | 6 and 12 months post-intervention
  A binary variable indicating whether the man reported having receptive anal intercourse in the past 90 days.
Insertive anal intercourse in the past 3 months | 6 and 12 months post-intervention
  A binary variable indicating whether the participant reported having insertive anal intercourse with a man in the past 90 days.
Proportion condom-protected intercourse in the past 3 months | 6 and 12 months post-intervention
  The denominator was the sum of reported anal and vaginal intercourse acts in the past 90 days and the numerator was the sum of condom-protected anal and vaginal intercourse act in the past 90 days.
Multiple sexual partners in the past 3 months | 6 and 12 months post-intervention
  Participants whose sum of anal and vaginal intercourse partners in the past 90 days was 2 or greater were coded as having multiple partners, and those who reported having 0 or 1 anal and vaginal intercourse partners in the past 90 days were coded as not having multiple partners.
Unprotected intercourse in the past 3 months | 6 and 12 months post-intervention
  A binary variable indicating whether the participants reported having vaginal or anal intercourse in the past 90 days without using a condom. It was constructed by subtracting the sum of the condom-protected anal and vaginal intercourse acts from the total number of anal and vaginal intercourse acts in the past 90 days. If the difference was one or greater the participant was coded as having unprotected intercourse; if the difference was zero or if the person reported no vaginal or anal intercourse in the past 90 days, the person was coded as not having unprotected intercourse.

CONTACTS AND LOCATIONS:
Overall Officials: John B Jemmott III, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Stevens R, Bernadini S, Jemmott JB. Social environment and sexual risk-taking among gay and transgender African American youth. Cult Health Sex. 2013;15(10):1148-61. doi: 10.1080/13691058.2013.809608. Epub 2013 Jul 26. PMID 23889233
- [Background] O'Leary A, Jemmott JB 3rd, Stevens R, Rutledge SE, Icard LD. Optimism and education buffer the effects of syndemic conditions on HIV status among African American men who have sex with men. AIDS Behav. 2014 Nov;18(11):2080-8. doi: 10.1007/s10461-014-0708-0. PMID 24705710
- [Result] Jemmott JB 3rd, Jemmott LS, O'Leary A, Icard LD, Rutledge SE, Stevens R, Hsu J, Stephens AJ. On the Efficacy and Mediation of a One-on-One HIV Risk-Reduction Intervention for African American Men Who Have Sex with Men: A Randomized Controlled Trial. AIDS Behav. 2015 Jul;19(7):1247-62. doi: 10.1007/s10461-014-0961-2. PMID 25449552
- [Derived] Zhang J, Jemmott JB 3rd, O'Leary A, Stevens R, Jemmott LS, Icard LD, Hsu J, Rutledge SE. Efficacy and Mediation of a Theory-Based Physical Activity Intervention for African American Men Who Have Sex with Men: A Randomized Controlled Trial. Ann Behav Med. 2017 Feb;51(1):106-116. doi: 10.1007/s12160-016-9832-6. PMID 27658914